CLINICAL TRIAL: NCT05852938
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study of BION-1301 in Adults With IgA Nephropathy (The BEYOND Study)
Brief Title: A Study of Zigakibart in Adults With IgA Nephropathy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFUB523A12301; CHK02-02 (Other: Chinook Therapeutics)
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-05

CONDITIONS: IgA Nephropathy; Immunoglobulin A Nephropathy
Keywords: Kidney Diseases; Kidney Diseases, Chronic; Urological Diseases; Glomerulonephritis; Glomerular Disease; Glomerulonephritis, IGA; Glomerulopathy; Immunoglobulin Disease
MeSH Terms: conditions — Glomerulonephritis, IGA; Kidney Diseases; Renal Insufficiency, Chronic; Urologic Diseases; Glomerulonephritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BION-1301 (Experimental): 600mg subcutaneous administration every 2 weeks for 104 weeks
  Interventions: Drug: BION-1301
- Placebo (Placebo Comparator): subcutaneous administration every 2 weeks for 104 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BION-1301 — BION-1301 Pre-Filled Syringe (PFS) 600mg subcutaneous administration every 2 weeks for 104 weeks.
  Other Names: Zigakibart
  Arms: BION-1301
Drug: Placebo — Placebo - PFS subcutaneous administration every 2 weeks for 104 weeks.
  Arms: Placebo

SUMMARY:
Safety and Efficacy of BION-1301 in Adults with IgA Nephropathy

DETAILED DESCRIPTION:
Approximately 330 participants with eGFR ≥ 30 mL/min/1.73m^2 and with biopsy-proven IgAN will be randomized to receive 600 mg Q2W BION-1301 or a matched placebo for 104 weeks. An additional exploratory cohort, not included in the primary analysis, will be comprised of approximately 20 participants (10 participants per arm) with biopsy-confirmed IgAN and eGFR of ≥ 20 to < 30 mL/min/1.73 m^2. The exploratory cohort will be randomized using the same schema as the primary cohort.

The primary objective of the study is to evaluate the effect of BION-1301 versus placebo on proteinuria in adults with IgA nephropathy.

Participants will have assessments of safety and efficacy for up to 2.5 years (134 weeks). To facilitate study participation over this time period, other visits may be remote (away from study site) for participants who elect to self-administer the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged ≥ 18 years at the time of signing the informed consent form (ICF) prior to initiation of any study specific activities/procedures.
* Biopsy-proven IgAN diagnosed within the past 10 years prior to Screening, that, in the opinion of the Investigator, is not due to secondary causes. A pseudonymized copy of the report must be available for review by the Sponsor or designee prior to randomization. If biopsy report within 10 years is not available, re-biopsy may be permitted upon discussion with the Sponsor.
* eGFR ≥ 30 mL/min/1.73m^2 at Screening based on the 2021 CKD-EPI equation.
* Total urine protein ≥ 1.0 g/day or UPCR ≥ 0.7 g/g (700 mg/g), as measured from an adequate 24-hour urine collection at Screening by a central laboratory.
* Stable on a maximally tolerated dose of angiotensin-converting enzyme inhibitors (ACEi) and/or angiotensin II receptor blockers (ARB) for at least 12 weeks prior to Screening unless intolerant to ACEi and ARB. May also be on a stable and well tolerated dose of sodium glucose cotransporter-2 inhibitors (SGLT2i), endothelin receptor antagonists (ERAs) and/or mineralocorticoid receptor antagonists (MRAs) for at least 12 weeks prior to Screening for the treatment of IgAN. Subjects are expected to stay on a stable dose of ACEi, ARB, SGLT2i, ERAs, and/or MRAs for the duration of the study.
* Screening weight of 45 to 150 kg.
* Men and women of childbearing potential (WOCBP; per Clinical Trials Facilitation and Coordination Group [CTFG] 2020) must agree to follow protocol-specified contraception guidance from Screening through approximately 5 half-lives (24 weeks) after the final dose of study drug. Use of hormonal contraceptive agents must have been initiated > 1 month prior to first dose of study drug.
* Provide written informed consent and be willing to comply with study visits and procedures.

Exclusion Criteria:

* Secondary forms of IgAN as determined by the Investigator, in the setting of systemic disorders, infections, autoimmune disorders or neoplasias.
* Diagnosis of IgA Vasculitis.
* Current or history of nephrotic syndrome.
* Average blood pressure > 150/90 mm Hg (systolic/diastolic) from 3 readings obtained at the initial Screening visit. If blood pressure is too high, the 3 readings may be repeated once within the Screening period if clinically appropriate as per the Investigator.
* Clinical suspicion of IgAN with rapidly progressive glomerulonephritis (RPGN) based on KDIGO guidelines
* Chronic Kidney Disease, either clinically suspected or based on biopsy, resulting from any condition or another glomerulopathy/podocytopathy other than IgAN.
* History of Type 1 Diabetes.
* Participants with Type 2 diabetes are excluded if any of the following are present:

  * Screening HbA1c (glycated hemoglobin) of > 8%.
  * Evidence of diabetic changes on kidney biopsy, performed for any reason.
  * History of diabetic microvascular disease (retinopathy, neuropathy, nephropathy) and/or macrovascular disease (atherosclerotic heart disease, peripheral vascular disease, cerebrovascular disease).
  * Unstable anti-diabetic regimen:
* Prior exposure to any therapy directed against APRIL.
* History of a previous severe allergic reaction with generalized urticaria, angioedema, or anaphylaxis, including a history of allergy or hypersensitivity to any component of BION-1301, or history of severe hypersensitivity reaction to any monoclonal antibody.
* Received an investigational new drug within 28 days or 5 half-lives, whichever is longer, prior to Screening.
* Received systemic corticosteroid therapy including budesonide (Tarpeyo/Kinpeygo) for > 14 days within 12 weeks prior to Screening.
* Use of systemic immunosuppressant medications.
* Any confirmed or suspected immunosuppressive or immune-deficient state, including but not limited to common variable immunodeficiency (CVID), HIV infection or asplenia, history of bone marrow or organ transplantation with exception of corneal transplants.
* Current severe infection requiring antimicrobials or history of recurrent, severe, infections as determined by the Investigator.
* Positive serology test for hepatitis A virus IgM antibodies (anti-HAV IgM), hepatitis B surface antigen (HBsAg), detectable hepatitis B virus (HBV) DNA, hepatitis C virus (HCV) antibodies (participants who completed treatment and are persistently antibody be allowed), or antibodies to HIV-1 and/or HIV-2 at Screening.
* Received a live vaccination within 12 weeks prior to Screening or plan to have a live vaccination within 6 months after the last dose of study drug.
* History of malignancy unless cancer free for at least 5 years or non-melanoma skin cancer that was completely resected. A participant with curatively treated cervical carcinoma in situ is eligible for the study. Participants with low-risk prostate cancer (i.e., Gleason score < 7 and prostate specific antigen < 10 ng/mL) are allowed.
* Pregnancy or breastfeeding or intent to become pregnant or to donate sperm during the study period and until 24 weeks after last dose.
* History or evidence of any other clinically significant disorder, condition, disease, or laboratory finding that, in the Investigator's assessment, would place the participant at unacceptable risk, limit compliance with study requirements, or confound interpretation of study results.
* IgG levels < 6 g/L at Screening.
* Participation in another interventional trial with an investigational agent/device is prohibited during the course of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2026-02-19 (Estimated); Study Completion 2028-06-07 (Estimated)

PRIMARY OUTCOMES:
Change in proteinuria (natural log UPCR) | 40 weeks or approximately 9 months
  The change in urine protein: creatinine ratio (UPCR) from baseline to Week 40.

SECONDARY OUTCOMES:
Annualized rate of change in eGFR | 104 weeks or approximately 2 years
  Annualized eGFR slope estimated over 104 weeks using the CKD-EPI 2021 creatinine equation
Change from baseline in eGFR | 104 weeks or approximately 2 years
  Change from Baseline to Week 104 in eGFR using the CKD-EPI 2021 creatinine equation
Effect of BION-1301 on specific clinical composite endpoints (30% eGFR reduction) | Baseline and Weeks 4, 12, 24, 40, 52, 64, 76, 88, and 104
  Percent of participants meeting the composite endpoint of experiencing at least 1 of the following during the study:
  * At least 30% reduction in eGFR sustained for at least 30 days
  * eGFR < 15 mL/min/1.73m^2, sustained for at least 30 days
  * Chronic dialysis, ≥ 30 days
  * Kidney transplantation
  * All-cause mortality
Effect of BION-1301 on specific clinical composite endpoints (40% eGFR reduction) | Baseline and Weeks 4, 12, 24, 40, 52, 64, 76, 88, and 104
  Percent of participants meeting the composite endpoint of experiencing at least 1 of the following during the study:
  * At least 40% reduction in eGFR sustained for at least 30 days
  * eGFR < 15 mL/min/1.73m^2, sustained for at least 30 days
  * Chronic dialysis, ≥ 30 days
  * Kidney transplantation
  * All-cause mortality
Percent Change in Proteinuria and Total Urine Protein | 40 weeks or approximately 9 months
  Percent of participants achieving reduction of proteinuria to < 1.0 g/day at Week 40 and a ≥ 25% decrease in total urine protein from Baseline

CONTACTS AND LOCATIONS:
Locations (191):
- United States (28):
  - University of Alabama at Birmingham: The Kirklin Clinic, Birmingham, Alabama
  - Nephrology Consultants, LLC, Huntsville, Alabama
  - University of California, San Francisco, San Francisco, California
  - Valiance Clinical Research, South Gate, California
  - University of Colorado Hospital, Aurora, Colorado
  - Denver Nephrology Research Division, Denver, Colorado
  - Vida Medical Centers - Pembroke Pines, Pembroke Pines, Florida
  - NorthShore University HealthSystem, Evanston, Illinois
  - Nephrology Associales of Northern Illinois and Indiana, Hinsdale, Illinois
  - Nephrology Associates of Northern Illinois and Indiana - 7836 W Jefferson Blvd, Fort Wayne, Indiana
  - University Of Iowa Hospitals And Clinics, Iowa City, Iowa
  - Intermed Consultants, Edina, Minnesota
  - Capital District Renal Physicians, Clifton Park, New York
  - Nephrology Associates PC - Flushing, Flushing, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Cincinnati College of Medicine - 231 Albert Sabin Way, Cincinnati, Ohio
  - Cleveland Clinic-9500 Euclid Ave, Cleveland, Ohio
  - OHSU - Oregon Clinical and Translational Research Institute, Portland, Oregon
  - Northeast Clinical Research Center, LLC, Bethlehem, Pennsylvania
  - Columbia Nephrology Associates , P.A. - Columbia, Columbia, South Carolina
  - Knoxville Kidney Center, PLLC - Frenova F1, Knoxville, Tennessee
  - Dallas Renal Group - 1411 N Beckley Ave, Dallas, Texas
  - Dallas Renal Group - Waxachie - 2460 N. I-35, Dallas, Texas
  - DaVita Clinical Research, El Paso, Texas
  - University of Texas MD Anderson Cancer Center-1155 Pressler, Houston, Texas
  - East Texas Nephrology Associates, Lufkin, Texas
  - Nephrology Associates of Northern Virginia-8501 Arlington Blvd, Fairfax, Virginia
  - Swedish Center for Comprehensive Care, Seattle, Washington
- Argentina (6):
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Catamarca, Catamarca Province
  - Novartis Investigative Site, Barracas, Ciudad Autónoma de BuenosAires
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Santa Fe, Santa Fe Province
  - Novartis Investigative Site, Buenos Aires
- Australia (8):
  - Novartis Investigative Site, Gosford, New South Wales
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Liverpool, New South Wales
  - Novartis Investigative Site, Penrith, New South Wales
  - Novartis Investigative Site, St Leonards, New South Wales
  - Novartis Investigative Site, Cairns North, Queensland
  - Novartis Investigative Site, Box Hill, Victoria
  - Novartis Investigative Site, St Albans, Victoria
- Belgium (6):
  - Novartis Investigative Site, Bonheiden, Antwerpen
  - Novartis Investigative Site, Ghent, Oost-Vlaanderen
  - Novartis Investigative Site, Roeselare, West-Vlaanderen
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Lodelinsart
  - Novartis Investigative Site, Woluwe-Saint-Lambert
- Brazil (8):
  - Novartis Investigative Site, Santana, Amapá
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Maringá, Paraná
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Joinville, Santa Catarina
  - Novartis Investigative Site, São Bernardo do Campo, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, São Paulo
- Canada (7):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, East York, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Montreal, Quebec
- China (21):
  - Novartis Investigative Site, Hefei, Anhui
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Foshan, Guangdong
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shenzhen, Guangdong
  - Novartis Investigative Site, Nanning, Guangxi
  - Novartis Investigative Site, Guiyang, Guizhou
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Nantong, Jiangsu
  - Novartis Investigative Site, Wuxi, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Jinan, Shandong
  - Novartis Investigative Site, Qingdao, Shandong
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Taiyuan, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Ürümqi, Xinjiang
  - Novartis Investigative Site, Wulumuji, Xinjiang
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Taizhou, Zhejiang
- Croatia (4):
  - Novartis Investigative Site, Zagreb, City of Zagreb
  - Novartis Investigative Site, Biškupec Zelinski
  - Novartis Investigative Site, Rijeka
  - Novartis Investigative Site, Vinkovci
- Novartis Investigative Site, Prague, Praha, Hlavní Mesto, Czechia
- France (5):
  - Novartis Investigative Site, Nîmes, Gard
  - Novartis Investigative Site, Lille, Nord
  - Novartis Investigative Site, Lyon, Rhône
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Paris
- Germany (7):
  - Novartis Investigative Site, Augsburg, Bavaria
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Mainz, Rhineland-Palatinate
  - Novartis Investigative Site, Trier, Rhineland-Palatinate
  - Novartis Investigative Site, Magdeburg, Saxony-Anhalt
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Essen
- Greece (6):
  - Novartis Investigative Site, Pátrai, Achaïa
  - Novartis Investigative Site, Athens, Attica
  - Novartis Investigative Site, Kalamaria, Thessaloniki
  - Novartis Investigative Site, Heralkion
  - Novartis Investigative Site, Ioannina
  - Novartis Investigative Site, Thessaloniki
- India (10):
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Chandigarh, Chandigarh
  - Novartis Investigative Site, Faridabad, Haryana
  - Novartis Investigative Site, Bengaluru, Karnataka
  - Novartis Investigative Site, Trivandrum, Kerala
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Vellore, Tamil Nadu
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, Dehradun
- Israel (6):
  - Novartis Investigative Site, Beersheba, Southern District
  - Novartis Investigative Site, Holon, Tel Aviv
  - Novartis Investigative Site, Ramat Gan, Tel Aviv
  - Novartis Investigative Site, Be’er Ya‘aqov
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (7):
  - Novartis Investigative Site, Bari, Apulia
  - Novartis Investigative Site, Foggia, Apulia
  - Novartis Investigative Site, Napoli, Campania
  - Novartis Investigative Site, Modena, Emilia-Romagna
  - Novartis Investigative Site, Trieste, Friuli Venezia Giulia
  - Novartis Investigative Site, Pavia, Lombardy
  - Novartis Investigative Site, Ranica, Lombardy
- Japan (18):
  - Novartis Investigative Site, Kasugai-Shi, Aiti
  - Novartis Investigative Site, Toyoake-shi, Aiti
  - Novartis Investigative Site, Urayasu-Shi, Chiba
  - Novartis Investigative Site, Sapporo, Hokkaidô
  - Novartis Investigative Site, Kitakyushu, Hukuoka
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kashihara, Nara
  - Novartis Investigative Site, Nara, Nara
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Bunkyo-Ku, Tokyo
  - Novartis Investigative Site, Hachioji-Shi, Tokyo
  - Novartis Investigative Site, Minato-Ku, Tokyo
  - Novartis Investigative Site, Shinjuku-Ku, Tokyo
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Niigata
  - Novartis Investigative Site, Okayama
  - Novartis Investigative Site, Tokyo
  - Novartis Investigative Site, Yufu-Shi, Ôita
- Malaysia (4):
  - Novartis Investigative Site, Kuantan, Pahang
  - Novartis Investigative Site, Sibu, Sarawak
  - Novartis Investigative Site, Kajang, Selangor
  - Novartis Investigative Site, Kuala Lumpur, WilayahPersekutuan KualaLumpur
- Mexico (6):
  - Novartis Investigative Site, Chihuahua, Chiapas
  - Novartis Investigative Site, Barrio Belisario Domínguez Secc, Mexico City
  - Novartis Investigative Site, Oaxaca, Mexico City
  - Novartis Investigative Site, Aguascalientes
  - Novartis Investigative Site, Chihuahua City
  - Novartis Investigative Site, Monterrey
- South Korea (9):
  - Novartis Investigative Site, Dongan-Gu, Anyang-Si, Gyeonggido
  - Novartis Investigative Site, Guri-si, Gyeonggido
  - Novartis Investigative Site, Uijeongbu-si, Gyeonggido
  - Novartis Investigative Site, Jongno-gu, Seoul Teugbyeolsi
  - Novartis Investigative Site, Seodaemun-gu, Seoul Teugbyeolsi
  - Novartis Investigative Site, Seongbuk-Gu, Seoul Teugbyeolsi
  - Novartis Investigative Site, Cheonan
  - Novartis Investigative Site, Daejeon
  - Novartis Investigative Site, Seoul
- Spain (7):
  - Novartis Investigative Site, Manises, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Girona
  - Novartis Investigative Site, Lleida
  - Novartis Investigative Site, Lugo
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Seville
- Taiwan (7):
  - Novartis Investigative Site, Keelung, Keelung
  - Novartis Investigative Site, Changhua County
  - Novartis Investigative Site, Hsinchu
  - Novartis Investigative Site, Hualien City
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Bornova, İzmir
  - Novartis Investigative Site, İzmit, Kocaeli
  - Novartis Investigative Site, Antalya
  - Novartis Investigative Site, Kayseri
- United Kingdom (6):
  - Novartis Investigative Site, Bristol, Bristol, City of
  - Novartis Investigative Site, Brighton, East Sussex
  - Novartis Investigative Site, Salford, Lancashire
  - Novartis Investigative Site, Leicester, Leicestershire
  - Novartis Investigative Site, London, London, City of
  - Novartis Investigative Site, Nottingham, Nottinghamshire

REFERENCES:
- [Derived] Kooienga L, Lo J, Lee EY, Kim SG, Thomas H, Workeneh B, Agha I, Song Y, Smith W, van Eenennaam H, Van Elsas A, Dulos J, Barratt J. Zigakibart demonstrates clinical safety and efficacy in a Phase 1/2 trial of healthy volunteers and patients with IgA nephropathy. Kidney Int. 2025 Sep;108(3):445-454. doi: 10.1016/j.kint.2025.05.006. Epub 2025 Jun 5. PMID 40482854
- [Derived] Ahmad SB, Jefferson JA. Targeting B Cells and Plasma Cells in Glomerular Disease. J Am Soc Nephrol. 2025 Jun 4;36(9):1844-1857. doi: 10.1681/ASN.0000000772. PMID 40465397
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639